CLINICAL TRIAL: NCT07291024
Title: Vagus Nerve Stimulation (VNS) Paired With Mobility Training For Gait Recovery After Chronic Ischemic Stroke With Integration Of Biomarker Assessment
Brief Title: A Study Of Vagus Nerve Stimulation (VNS) With Mobility Training For Gait Recovery After Chronic Ischemic Stroke
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Mayo Clinic (Other)
Responsible Party: Principal Investigator, Rushna Ali, Principal Investigator, Mayo Clinic
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 25-008515
Record Dates: First submitted 2025-12-05; First posted 2025-12-18 (Actual); Last update posted 2025-12-18 (Actual); Status verified 2025-12

CONDITIONS: Ischemic Stroke
MeSH Terms: conditions — Ischemic Stroke | interventions — Vagus Nerve Stimulation

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Chronic ischemic stroke (Experimental): Participants with chronic ischemic stroke will be treated with a combination of vagus nerve stimulation and mobility training.
  Interventions: Other: Vagus nerve stimulation (VNS) paired with mobility training

INTERVENTIONS:
Other: Vagus nerve stimulation (VNS) paired with mobility training — Participants will complete a 6-week in-clinic therapy phase (3 sessions per week), where a physical therapist will lead mobility training with VNS delivered via a handheld magnet. This will be followed by a 6-week at-home phase where participants continue daily exercises and VNS use, supported by weekly video calls to review at home rehabilitation activity and wearable activity monitors for remote monitoring.

SUMMARY:
The purpose of this study is to evaluate the safety, feasibility, and efficacy of vagus nerve stimulation (VNS) paired with mobility training to improve lower extremity function and gait in individuals with chronic ischemic stroke.

ELIGIBILITY:
Inclusion Criteria:

* Age ≥ 18 years
* Ischemic stroke ≥6 months prior to enrollment.
* Post-stroke lower extremity impairment defined as gait velocity of less than 0.8 m/s on a 10-meter walk test
* Provision of informed consent

Exclusion Criteria:

* Intracerebral Hemorrhage
* Active or prior psychosis or substance abuse within two years.
* Pre-stroke modified Rankin Scale (mRS) 3-5.
* Unable to participate in in-clinic rehabilitation.
* Preexisting neurological disorders affecting gait and mobility, such as Parkinson's disease, Amyotrophic Lateral Sclerosis (ALS), Multiple Sclerosis (MS), dementia, major head trauma.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Estimated)
Dates: Start 2026-01-01 (Estimated); Primary Completion 2029-01-01 (Estimated); Study Completion 2029-01-01 (Estimated)

PRIMARY OUTCOMES:
Number of serious adverse events related to vagus nerve stimulation or therapy | 1 year
  Total number of serious adverse events reported related to vagus nerve stimulation (VNS) or mobility training
Number of participants to complete the study | 1 year
  Total number of participants to complete a minimum of 18 therapy sessions
Change in Instrumented Gait Assessment score | Baseline, 12 months
  Gait speed is calculated as the predetermined distance divided by the time to walk that distance, reported in meters per second (m/s). Improvement in gait velocity is ≥0.05 m/s .

CONTACTS AND LOCATIONS:
Overall Officials: Rushna Ali, MD, Principal Investigator — Mayo Clinic; Muhib Khan, MD, MBBS, Principal Investigator — Mayo Clinic
Locations (1):
- Mayo Clinic in Rochester, Rochester, Minnesota, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- See also: Mayo Clinic Clinical Trials — https://www.mayo.edu/research/clinical-trials